CLINICAL TRIAL: NCT06720077
Title: Effect of Acupressure in The Management of Postmenopausal Constipation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samar Gamal Mohamed Gab Allah, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004870
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — Acupressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupressure + diaphragmatic breathing exercises + general bowel care advise (Experimental): It consisted of 30 postmenopausal women. Each of them received acupressure on the (san jio 6/ stomach 25/ spleen 15/ joining vally " large intestine 4 ") acupoints, 1 minute for each point with 3 repetitions on both sides (about 30 minutes as total time), 3 times per week in addition to diaphragmatic breathing exercises for 15 minutes and general bowel care advise, for 6 weeks.
  Interventions: Other: Acupressure; Other: Diaphragmatic breathing exercises; Other: General bowel care advise
- diaphragmatic breathing exercises + general bowel care advise (Active Comparator): It consisted of 30 postmenopausal women who performed diaphragmatic breathing exercises for 15 minutes 3 times per week in addition to general bowel care advice only, for 6 weeks.
  Interventions: Other: Diaphragmatic breathing exercises; Other: General bowel care advise

INTERVENTIONS:
Other: Acupressure — It will be applied for the experimental group only. Before starting the first treatment session, the participants will be instructed briefly about the nature of the treatment to gain their confidence and cooperation. Each participant in this group will be asked to lie in supine position and the acupressure will be applied by using the therapist's fingers on the following acupoints (san jio 6/ spleen 15/ stomach 25/ joining vally " intestine 4") 1 minute for each point with 3 repetitions on both sides (about 30 minutes as total time), 3 times per week for 6 weeks.
  Arms: acupressure + diaphragmatic breathing exercises + general bowel care advise
Other: Diaphragmatic breathing exercises — A modified exercise will be used to achieve normal diaphragmatic breathing while the woman is lying on her back, with one hand placed on her abdomen and the other on her thorax. She will then be instructed to breathe in deeply, slowly, and gradually for 4 seconds, hold the air for 2 seconds, and exhale slowly through pursed lips for 6 seconds. Three series of ten repetitions will be completed with rest in between; the woman will be advised to rest longer if she feels dizzy or lightheaded. The patient will ensure the exercise is performed successfully if the hand placed on the abdomen shows greater mobility compared to minimal or no mobility of the hand on the thorax. From that point, the series of repetitions will begin.
Other: General bowel care advise — All women in both groups will receive bowel care advice, including encouraging fiber intake (20-35 g/day) from sources like whole grains, fruits, vegetables, and legumes, with a focus on soluble fiber. They will be advised to limit meat, dairy, and low-fiber foods and avoid caffeine-containing products like chocolate and coffee. Adequate hydration (1.5-2.0 L/day) with water or juices will be recommended, along with daily exercise, such as 20-30 minutes of walking. Proper toilet posture will be emphasized, including sitting with knees higher than hips (using a stool if needed), leaning forward, placing elbows on knees, relaxing, and maintaining a straight spine.

SUMMARY:
This study was conducted to investigate the effect of acupressure in the management of constipation in postmenopausal women.

DETAILED DESCRIPTION:
Constipation is prevalent in menopause, affecting 4-29% of women globally, and can lead to serious complications like hemorrhoids, anal fissures, and colorectal cancer. While laxatives can help, long-term use may cause dependency and side effects. Alternative therapies are needed.

Deep breathing, particularly diaphragmatic breathing, may improve constipation by activating the parasympathetic system and promoting relaxation. Acupressure has also shown potential in managing constipation by stimulating intestinal activity, improving blood circulation, and regulating Qi flow.

Despite existing studies on acupressure and constipation, no research has specifically examined its effect on postmenopausal women. This study aims to investigate acupressure's impact on functional constipation in this population, offering potential insights for non-pharmacological management.

ELIGIBILITY:
Inclusion Criteria:

1. Sixty postmenopausal women who were clinically diagnosed as having functional constipation after menopause (at least one year after the stoppage of the last menstrual cycle)
2. Their ages ranged from 50 to 60 years old.
3. Their body mass index didn't exceed 30 kg/m2.
4. All of them should have at least two criteria of Rome III diagnostic criteria of constipation.
5. They should stop laxatives intake during the treatment program.

Exclusion Criteria:

1. Irritable bowel syndrome or anal fissures.
2. Genital organ prolapse as rectocele.
3. Any neurological diseases, spinal diseases or spinal deformities.
4. History of bowel surgery.
5. Congenital anorectal malformation, stoma in situ.
6. Diabetes mellitus and sever distal venous insufficiency.
7. Skin eruption at the site of stimulation.
8. Implanted pacemaker or defibrillator.
9. Metalic implant in lower limb.
10. Recent surgery at the lower limb.
11. Peripheral neuropathy and neurological disorders.
12. Psychological distress.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-07 (Estimated); Primary Completion 2025-02-20 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Patient Assessment of Constipation Symptom (PAC - SYM) | 6 weeks
  It is a reliable and valid tool to measure the patient's perspective constipation symptoms in terms of frequency and severity, It is a 12- item that is divided into three symptom subscales: abdominal (four items); rectal (three items); and stool (five items). Items are scored on 5-point Like scales, with scores ranging from 0 to 4 (0 = 'symptom absent', 1 = 'mild', 2 = 'moderate', 3 = 'severe' and 4 = 'very severe'). A mean total score in the range of 0-4 is generated by dividing the total score by the number of questions completed; the lower the total score, the lower the symptom burden.
Patient Assessment of Constipation quality of life (PAC - QOL) | 6 weeks
  The PAC-QOL questionnaire is used to evaluate the quality of life of patients having constipation. It is a brief but comprehensive tool which evaluates constipation through daily individual health assessment and functioning. This questionnaire consists of 28 self-reported items which sub-categorized to 4 items on physical discomfort, 8 items on psychosocial discomfort, 5 items on treatment satisfaction, and finally 11 items on worries and discomfort. Lower scores indicate higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Azza Barmoud Nashed Kassab, PhD, Study Chair — Professor, Cairo university
Locations (1):
- Faculty of physical therapy, Cairo University, Giza, Egypt